CLINICAL TRIAL: NCT00292851
Title: Repeatability and Validity of Measurements in Blown Nasal Secretion in Patients With Rhinosinusitis
Brief Title: Blown Nasal Secretion Measurements in Rhinosinusitis: Repeatability and Validity Compared to Nasal Lavage
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Dr. Frederick Hargreave, St. Joseph's Healthcare Hamilton/McMaster University
Other Study IDs: RP#02-2075
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To process blown nasal secretions from subjects with rhinosinusitis and to obtain a specimen by nasal lavage. To investigate the reliability and validity of the measurements we will determine their repeatability and compare them with those of nasal lavage in the same subjects.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from rhinitis with our without sinusitis

Exclusion Criteria:

* unable to provide blown nasal sample

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with rhinitis
Sampling Method: Probability Sample
Enrollment: 15
Dates: Start 2004-07; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E Hargreave, MD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada